CLINICAL TRIAL: NCT01123499
Title: Collection of Peripheral Blood Stem Cells Using G-CSF and Plerixafor in Healthy Volunteers
Brief Title: Collection of Peripheral Blood Stem Cells Using G-CSF and Plerixafor in Normal Volunteers
Status: Terminated | Type: Observational
Why Stopped: Slow/Insufficient accrual
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 100095; 10-I-0095
Record Dates: First submitted 2010-05-13; First posted 2010-05-14 (Estimated); Last update posted 2022-05-06 (Actual); Status verified 2021-05

CONDITIONS: Normal Physiology
Keywords: G-CSF; Plerixafor; Mozobil; Apheresis; Healthy Volunteer; Natural History; HV

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood

GROUPS / COHORTS (1):
- Healthy Volunteers: Any healthy volunteers that are eligible to donate blood.

SUMMARY:
Background:

* Many treatments for immune system disorders involve the use of stem cells that have been collected from blood marrow. To obtain these stem cells without surgery, individuals receive granulocyte colony-stimulating factor (G-CSF) to encourage the production of stem cells that can be collected through blood donations. However, not all patients or normal donors respond to G-CSF alone.
* Plerixafor, recently approved by the Food and Drug Administration, is different from G-CSF but also allows stem cells to be collected from donated blood. However, more research is needed on the quality and viability of the stem cells collected after using both G-CSF and plerixafor.

Objectives:

- To collect and study the blood cells produced after treatment with G-CSF and plerixafor in healthy volunteers.

Eligibility:

- Healthy volunteers between 18 and 65 years of age who are eligible to donate blood.

Design:

* Participants will be screened with a medical history, physical examination, and initial blood tests.
* At the start of the study cycle, participants will receive daily morning injections of G-CSF for 5 days. These may be given at the clinical center or by the participant after teaching, depending on the participant s preference.
* On the morning of Day 4, participants will visit the clinical center to provide a blood sample after the injection. On the evening of Day 4, participants will receive an injection of plerixafor.
* Participants will have the final injection of G-CSF on the morning of Day 5, and will provide another blood sample.
* On Day 5, participants will have apheresis to separate the stem cells from the rest of the blood. The apheresis may take up to 5 hours to complete.
* The study will end after a follow-up phone call 7 to 14 days after the apheresis procedure.

DETAILED DESCRIPTION:
Hematopoietic stem cells that have been mobilized from the bone marrow into the peripheral circulation are readily collected by apheresis, and may be used for several purposes. They are used for allogeneic and autologous transplantation and are often manipulated in various ways depending on the goal of the transplant. Gene therapy for immunodeficiencies relies on the collection of these cells.

Traditionally, mobilization has been done using granulocyte colony stimulating factor (G-CSF). However not all patients or normal donors respond to GCSF alone. Plerixafor, a recently Food and Drug Administration (FDA) approved drug, has a unique mode of action distinct from that of GCSF, but also results in mobilization of peripheral blood progenitors into the circulation, allowing their collection by standard apheresis. The quality of these cells for transduction using viral vectors in anticipation of gene therapy uses has not been thoroughly assessed, and there are theoretical considerations why vectors that use various envelopes for cell binding may be affected by the use of this CXCR4 antagonist. In order to be able to assess the transduction and engraftment of these cells in murine models, we will perform collection and mobilization on 5 healthy volunteers at the NIH Clinical Center using the FDA approved medications G-CSF and plerixafor.

ELIGIBILITY:
* INCLUSION CRITERIA:

To be eligible to participate in this study, a subject must satisfy all of the following criteria:

1. The subject must be a healthy adult aged 18-65 years, and weighing at least 50 kg.

2, The subject must have normal renal function (creatinine <1.5 mg/dL; <1 plus proteinuria); normal hepatic function (bilirubin < 1.5 mg/dL); normal hematologic function (WBC greater than or equal to 2500/mm(3); granulocytes greater than or equal to 1200/mm(3); platelets greater than or equal to 120,000; hematocrit greater than or equal to 38).

3. A female of childbearing potential may be entered if she is using 1 or 2 forms of effective contraception (depending on the type of contraception), and has a negative serum pregnancy test within 1 week of beginning G-CSF administration. She must continue with the effective contraception 3 months after receiving plerixafor

4. The subject must be willing to allow blood cell samples to be stored.

EXCLUSION CRITERIA:

A subject will be ineligible to participate in this study if any of the following criteria are met:

1. The subject has a temperature > 38 degrees Celsius, or WBC > 9000/mm(3).
2. A female who is pregnant or lactating as determined by history and/or pregnancy test.
3. The subject has a history of vasculitis, uncontrolled hypertension, or symptomatic coronary artery disease, or similar disorders.
4. The subject has a positive test result for any of the following: human immunodeficiency virus (HIV) I & II antibody, hepatitis C virus (HCV) antibody, hepatitis B soluble antigen (HBSAg), or the rapid plasma reagin (RPR) test for syphilis.
5. The subject lacks peripheral venous access in arm veins adequate for apheresis.
6. The subject is currently participating in other research studies.
7. The subject may be excluded at the discretion of the Principal Investigator (PI).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Any healthy volunteers that are eligible to donate blood.@@@@@@
Sampling Method: Non-Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2016-10-06 (Actual); Primary Completion 2017-01-27 (Actual); Study Completion 2022-04-28 (Actual)

PRIMARY OUTCOMES:
Apheresis | Time of Apheresis
  To collect cells from normal volunteers using both G-CSF and plerixafor, to be able to use these in various research applications.

SECONDARY OUTCOMES:
Apheresis | 6 months after collect of cells
  To characterize the grafts obtained from normal donors using G-CSF and plerixafor and to compare these grafts to historical grafts collected using G-CSF alone.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth M Kang, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Levesque JP, Hendy J, Takamatsu Y, Simmons PJ, Bendall LJ. Disruption of the CXCR4/CXCL12 chemotactic interaction during hematopoietic stem cell mobilization induced by GCSF or cyclophosphamide. J Clin Invest. 2003 Jan;111(2):187-96. doi: 10.1172/JCI15994. PMID 12531874
- [Background] Flomenberg N, Devine SM, Dipersio JF, Liesveld JL, McCarty JM, Rowley SD, Vesole DH, Badel K, Calandra G. The use of AMD3100 plus G-CSF for autologous hematopoietic progenitor cell mobilization is superior to G-CSF alone. Blood. 2005 Sep 1;106(5):1867-74. doi: 10.1182/blood-2005-02-0468. Epub 2005 May 12. PMID 15890685
- [Background] Liles WC, Broxmeyer HE, Rodger E, Wood B, Hubel K, Cooper S, Hangoc G, Bridger GJ, Henson GW, Calandra G, Dale DC. Mobilization of hematopoietic progenitor cells in healthy volunteers by AMD3100, a CXCR4 antagonist. Blood. 2003 Oct 15;102(8):2728-30. doi: 10.1182/blood-2003-02-0663. Epub 2003 Jul 10. PMID 12855591
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2010-I-0095.html